CLINICAL TRIAL: NCT02710435
Title: REDUCER-I: An Observational Study of the Neovasc Reducer™ System
Status: Active, not recruiting | Type: Observational
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 022-REDUCLN-001
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Angina Pectoris; Angina Pectoris, Stable; Chronic Stable Angina
Keywords: Coronary Sinus; Reducer; Refractory Angina; Angina Pectoris; Angina Pectoris, Stable; Chronic Stable Angina; Persistent Angina; Neovasc Reducer System; Refractory Angina Pectoris; Coronary Sinus Narrowing; Reversible Ischemic Heart Disease; Chronic Angina; End Stage Angina; Coronary Sinus Reduction; Coronary Sinus Reducer; Chronic Refractory Angina; Chronic Refractory Angina Pectoris
MeSH Terms: conditions — Angina Pectoris; Angina, Stable

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Arm 1 - Prospective: Includes eligible subjects in the prospective arm who undergo baseline testing followed by the Reducer System implant procedure
  Arm 1 has been closed to enrollment-March 2023
  Interventions: Device: Reducer System
- Arm 2 - COSIRA: Includes subjects who were previously enrolled and treated with the Reducer System during the COSIRA study and agree to participate in this long term follow up study
  Interventions: Device: Reducer System
- Arm 3 - CE Mark: Includes subjects who received a Reducer System under CE Mark (unrelated to the COSIRA study), and agree to participate in this long term follow up study
  Arm 3 has been closed to enrollment-June 2017
  Interventions: Device: Reducer System

INTERVENTIONS:
Device: Reducer System — An aid in the management of chronic refractory angina pectoris
  Other Names: Reducer

SUMMARY:
The purpose of this study is to collect long term data of the Reducer System in subjects with refractory angina pectoris.

DETAILED DESCRIPTION:
This study is a multicenter, multi-country three-arm prospective and retrospective investigation in up to 400 subjects conducted at a maximum of 40 investigational centers. Arm 1 will include eligible prospective subjects. Arm 2 will include subjects who were previously enrolled and treated with the Reducer during the COSIRA (Coronary Sinus Reducer for Treatment of Refractory Angina) study. Arm 3 will include subjects who received a Reducer under CE Mark (unrelated to the COSIRA study).

ELIGIBILITY:
Inclusion Criteria - ALL Arms:

* Subject has been informed about the study and provides written informed consent prior to enrollment
* Subject is willing to comply with specified follow-up evaluations

Inclusion Criteria - Arm 1:

* Symptomatic Coronary Artery Disease (CAD) with chronic refractory angina pectoris despite attempted optimal medical therapy
* Subject has limited treatment options for revascularization by Coronary Artery Bypass Grafting (CABG) or by Percutaneous Coronary Intervention (PCI)
* Evidence of reversible myocardial ischemia
* Left Ventricular ejection fraction (LVEF) greater than or equal to 30%
* Male or non-pregnant female

Inclusion Criteria - Arm 2:

* Subjects previously implanted in the Reducer (treatment) arm of the COSIRA study

Inclusion Criteria - Arm 3:

* Subjects in whom the Reducer was implanted under CE Mark (unrelated to the COSIRA study), prior to enrollment in the Reducer-I study

Exclusion Criteria - Arm 1:

* Acute coronary syndrome within three months prior to enrollment
* Recent successful revascularization by PCI or CABG within six months prior to enrollment
* Recent unsuccessful PCI (no relief from symptoms) within 30 days prior to enrollment
* Unstable angina (recent onset angina, crescendo angina, or rest angina with electrocardiogram [ECG] changes) during the 30 days prior to enrollment
* Decompensated congestive heart failure (CHF) or hospitalization due to CHF during the three months prior to enrollment
* Severe chronic obstructive pulmonary disease (COPD) as indicated by a forced expiratory volume in one second that is less than 55% of the predicted value
* Subject cannot undergo exercise tolerance test
* Subject cannot undergo 6-minute walk test
* Severe valvular heart disease
* Subject with pacemaker electrode in the coronary sinus (CS)
* Subject with recent placement of a new pacemaker or defibrillator electrode in the right atrium within 3 months prior to enrollment.
* Subject having undergone tricuspid valve replacement or repair
* Chronic renal failure (serum creatinine >2 mg/dL), including subjects on chronic hemodialysis
* Moribund subjects, or subjects with comorbidities limiting life expectancy to less than one year
* Known severe reaction to required procedural medications
* Known allergy to stainless steel or nickel
* Magnetic Resonance Imaging (MRI) planned within 8 weeks after Reducer implantation
* Currently enrolled in another device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints

Angiographic Exclusion:

* Mean right atrial pressure greater than 15mmHg
* Subject with anomalous or abnormal CS anatomy (e.g., tortuosity, aberrant branch, persistent left superior vena cava [SVC])
* CS diameter at the site of planned Reducer implantation less than 9.5 mm or greater than 13 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with refractory angina pectoris who demonstrate objective evidence of reversible myocardial ischemia, who have limited or no options for revascularization, or subjects who have received the Reducer in the COSIRA study, or under CE Mark prior to the REDUCER-I study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-03; Primary Completion 2023-11 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in Canadian Cardiovascular Society (CCS) Grade | 6 Months
  The percentage of subjects who experience improvement in their angina symptoms defined as a reduction in CCS grade, at 6 months as compared to baseline
Rate of Occurrence of Device and/or Procedure Related Peri-Procedural Serious Adverse Events (SAE)s | 30 days post implant
  The rate of occurrence of device and / or procedure-related periprocedural SAEs defined as a composite of death, Myocardial Infarction (MI), cardiac tamponade, clinically-driven re-dilation of a Reducer, life-threatening arrhythmias (Ventricular Tachycardia (VT) or Ventricular Fibrillation (VF)), and respiratory failure through 30 days post-implant
Occurrence of Major Adverse Cardiac Events (MACE) | 30 days post implant
  Major Adverse Cardiac Events (MACE): a composite of cardiac death, major stroke, and MI through 30-days post-implant

SECONDARY OUTCOMES:
Reduction in Canadian Cardiovascular Society (CCS) Grade | 12 months and annually through 5 years
  The percentage of subjects who experience improvement in their angina symptoms defined as a reduction in CCS grade at 12 months and annually through 5 years post implant as compared to baseline
Occurrence of Major Adverse Cardiac Events (MACE) | 6 months, 12 months, and annually through 5 years
  Major Adverse Cardiac Events (MACE): a composite of cardiac death, major stroke, and MI at 6 months, 12 months and annually through 5 years post implant

OTHER OUTCOMES:
Change in Exercise Tolerance Test (ETT) Parameters | 6 and 12 months
  The change in ETT parameters at 6 and 12 months post implant as compared to baseline: Total exercise duration (min), Time to 1mm ST-Segment Depression (min), METs, Double Product by ETT
Improvement in Quality of Life (QoL | 6 months, 12 months, and annually through 5 years
  Improvement in QoL scores at 6 months, 12 months and annually through 5 years post implant as compared to baseline
Reduction in Emergency Department Visits | 12 months
  Reduction in documented Emergency Department visits due to angina episodes at 12 months post implant as compared to 12 months prior to implantation of the Reducer
Reduction in Angina Medication | 6 months, 12 months, and annually through 5 years
  Reduction in angina medication use at 6 months, 12 months and annually through 5 years post implant as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, Principal Investigator — ZNA Middelheim Hospital
Locations (25):
- University of Graz, Graz, Austria
- Belgium (2):
  - ZNA Middelheim Hospital, Antwerp
  - Zienkenhuis Oost-Limburg, Genk
- France (2):
  - University Hospital of Brest, Brest
  - Institut Coeur Poumon, Lille
- Germany (6):
  - Kerckhoff Klinik, Bad Nauheim
  - Dresden University, Dresden
  - Contilia Heart and Vascular Centre, Elisabeth Krankenhaus Essen, Klinik fϋr Kardiologie und Angiologie, Essen
  - University Heart Center Freiburg - Bad Krozingen, Freiburg im Breisgau
  - University Giessen, Giessen
  - University Heart Center Hamburg, Hamburg
- Italy (2):
  - San Raffaele Hospital, Milan
  - Bolognini General Hospital, Seriate
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - UMC Utrecht, Utrecht
- Hospital Clinico San Carlos, Madrid, Spain
- Switzerland (4):
  - University Hospital Basel, Basel
  - HFR Fribourg/University of Fribourg, Fribourg
  - Hopitaux Universitaires Geneve (HUG), Geneva
  - Istituto Cardiocentro Ticino, Lugano
- United Kingdom (5):
  - Bradford Royal Infirmary, Bradford
  - Royal Infirmary of Edinburgh, Edinburgh
  - St. Thomas Hospital, London
  - King's College Hospital, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banai S, Ben Muvhar S, Parikh KH, Medina A, Sievert H, Seth A, Tsehori J, Paz Y, Sheinfeld A, Keren G. Coronary sinus reducer stent for the treatment of chronic refractory angina pectoris: a prospective, open-label, multicenter, safety feasibility first-in-man study. J Am Coll Cardiol. 2007 May 1;49(17):1783-9. doi: 10.1016/j.jacc.2007.01.061. PMID 17466229
- [Background] Banai S, Verheye S, Jolicoeur EM. A device to narrow the coronary sinus for angina. N Engl J Med. 2015 May 14;372(20):1967-8. doi: 10.1056/NEJMc1503672. No abstract available. PMID 25970058
- [Background] Verheye S, Jolicoeur EM, Behan MW, Pettersson T, Sainsbury P, Hill J, Vrolix M, Agostoni P, Engstrom T, Labinaz M, de Silva R, Schwartz M, Meyten N, Uren NG, Doucet S, Tanguay JF, Lindsay S, Henry TD, White CJ, Edelman ER, Banai S. Efficacy of a device to narrow the coronary sinus in refractory angina. N Engl J Med. 2015 Feb 5;372(6):519-27. doi: 10.1056/NEJMoa1402556. PMID 25651246
- [Background] Konigstein M, Verheye S, Jolicoeur EM, Banai S. Narrowing of the Coronary Sinus: A Device-Based Therapy for Persistent Angina Pectoris. Cardiol Rev. 2016 Sep-Oct;24(5):238-43. doi: 10.1097/CRD.0000000000000101. PMID 26886464
- [Background] Abawi M, Nijhoff F, Stella PR, Voskuil M, Benedetto D, Doevendans PA, Agostoni P. Safety and efficacy of a device to narrow the coronary sinus for the treatment of refractory angina: A single-centre real-world experience. Neth Heart J. 2016 Sep;24(9):544-51. doi: 10.1007/s12471-016-0862-2. PMID 27299456
- [Background] Konigstein M, Meyten N, Verheye S, Schwartz M, Banai S. Transcatheter treatment for refractory angina with the Coronary Sinus Reducer. EuroIntervention. 2014 Feb;9(10):1158-64. doi: 10.4244/EIJV9I10A196. PMID 24561732
- [Background] Verheye S, Agostoni P, Giannini F, Hill JM, Jensen C, Lindsay S, Stella PR, Redwood S, Banai S, Konigstein M. Coronary sinus narrowing for the treatment of refractory angina: a multicentre prospective open-label clinical study (the REDUCER-I study). EuroIntervention. 2021 Sep 20;17(7):561-568. doi: 10.4244/EIJ-D-20-00873. PMID 33319762
- See also: Company product webpage — https://shockwavemedical.com/clinicians/international/coronary/coronary-sinus-reduction/